CLINICAL TRIAL: NCT02803996
Title: Pharmacokinetics of Single and Multiple Escalating Doses of Aramchol Administered Under Fed Conditions in Healthy Chinese Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Galmed Pharmaceuticals Ltd (Industry)
Collaborators: WCCT Global (Industry); Alpha IRB (Unknown); Analyst Research Laboratories (Other); Kramer Consulting, LLC (Other); Diamond Pharma Services Regulatory Affairs Consultancy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple
Other Study IDs: Aramchol 015
Record Dates: First submitted 2016-06-07; First posted 2016-06-17 (Estimated); Last update posted 2016-12-21 (Estimated); Status verified 2016-12

CONDITIONS: Healthy Volunteers
MeSH Terms: interventions — aramchol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Part A- Single Dose- 400 mg Aramchol (Active Comparator): Part A: Subjects will receive a single dose of 400 mg Aramchol, 600 mg Aramchol or placebo.
  Interventions: Drug: Aramchol
- Part A- Single Dose- 600 mg Aramchol (Active Comparator): Part A: Subjects will receive a single dose of 400 mg Aramchol, 600 mg Aramchol or placebo.
  Interventions: Drug: Aramchol
- Part A-Single Dose-Placebo (Placebo Comparator): Part A: Subjects will receive a single dose of 400 mg Aramchol, 600 mg Aramchol or placebo.
  Interventions: Drug: Placebo
- Part B-Multiple Dose-400 mg Aramchol (Active Comparator): Part B: Subjects will receive multiple doses of 400 mg Aramchol, 600 mg Aramchol or placebo tablets for 10 consecutive days.
  Interventions: Drug: Aramchol
- Part B-Multiple Dose-600 mg Aramchol (Active Comparator): Part B: Subjects will receive multiple doses of 400 mg Aramchol, 600 mg Aramchol or placebo tablets for 10 consecutive days.
  Interventions: Drug: Aramchol
- Part B-Multiple Dose-Placebo (Placebo Comparator): Part B: Subjects will receive multiple doses of 400 mg Aramchol, 600 mg Aramchol or placebo tablets for 10 consecutive days.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aramchol — Part A: Aramchol oral tablets at 400 mg or 600 mg single dose Part B: Aramchol oral tablets at 400 mg or 600 mg multiple dose for 10 consecutive days.
  Arms: Part A- Single Dose- 400 mg Aramchol; Part A- Single Dose- 600 mg Aramchol; Part B-Multiple Dose-400 mg Aramchol; Part B-Multiple Dose-600 mg Aramchol
Drug: Placebo — Part A: Placebo oral tablets single dose Part B: Placebo oral tablets multiple dose for 10 consecutive days.
  Arms: Part A-Single Dose-Placebo; Part B-Multiple Dose-Placebo

SUMMARY:
This is a single-site, randomized, double-blind, double dummy, placebo-controlled single and multiple doses study of Aramchol in healthy Chinese volunteers. The subject population that was enrolled for Aramchol 004 was not specifically designed to understand the PK profile of Aramchol in subjects of Chinese descent. Therefore, this study (Aramchol 015) has been undertaken to ascertain the PK profile of Aramchol following single and multiple doses in a Chinese population under fed conditions utilizing the light breakfast from Aramchol 004.

This study will consist of two parts and the subjects will be assigned to two parts.

In each part of the study, subjects will be enrolled in the study within 28 days of screening.

DETAILED DESCRIPTION:
In each part of the study, subjects will be enrolled in the study within 28 days of screening. The study will consist of two parts, and the subjects will be assigned as follows: Part A- single escalating doses This part of the study is a single-site, randomized, double-blind, double dummy, placebo-controlled single-dose study of Aramchol in healthy Chinese volunteers. The purpose of Part A is to evaluate the PK, safety and tolerability of Aramchol tablets at single doses of either 400 mg or 600 mg.

Thirty-two (32) subjects will participate in this part of the study and will be randomized to receive a single-dose of 400 mg Aramchol, 600 mg Aramchol, or Placebo. Drug administration will be preceded by a light breakfast consumed within 1 hour prior to dosing. All drugs will be administered by the study staff. In order to maintain blinding, all subjects will receive two tablets on each dosing, according to the following administrations:

* Cohort A: 1 x 200 mg Placebo tablet + 1 x 400 mg Aramchol tablet (12 subjects)
* Cohort B: 1 x 200 mg Aramchol tablet + 1 x 400 mg Aramchol tablet (12 subjects)
* Cohort C: 1 x 200mg Placebo tablet + 1 x 400 mg Placebo tablet (8 subjects) Subjects will be admitted in-house in the evening before the first study drug administration (Day 0) and will remain in-house for 36 hours after dosing. Blood samples for Aramchol concentrations will be drawn for 36 hours at designated time points as described below. Additional ambulatory samples will be collected at 48, 72, 96, and 144 hours postdose. Subjects will be continuously monitored for safety. An End-of Study/Safety Follow-up visit will take place on the last PK sampling day, ie, 144 hours after the last dose administration.

If the PK profile from Part A is similar to the existing PK data in non- Chinese subjects, then the study may be stopped. If the PK profile is different, then Part B of the study may be performed.

Part B- multiple escalating doses Part B of the study is a single-site, randomized, double-blind, doubledummy, placebo-controlled multiple-dose study of Aramchol in healthy Chinese volunteers. The purpose of this part is to evaluate the PK, safety and tolerability of Aramchol tablets at multiple administrations of two different doses. Thirty-two (32) subjects will participate in this part of the study and will be equally randomized to receive 400 mg Aramchol, 600 mg Aramchol, or Placebo for 10 consecutive days. Screening for Part B may begin during PK analysis of Part A. Part A subjects can enroll into Part B with sponsor approval. Drug administration will be preceded by a light breakfast consumed within 1 hour prior to dosing. All drugs will be administered by the study staff. In order to maintain blinding, all subjects will receive two tablets on each dosing, according to the following administrations:

* Cohort D: 1 x 200 mg Placebo tablet + 1 x 400 mg Aramchol tablet (12 subjects)
* Cohort E: 1 x 200 mg Aramchol tablet + 1 x 400 mg Aramchol tablet (12 subjects)
* Cohort F: 1 x 200 mg Placebo tablet + 1 x 400 mg Placebo tablet (8 subjects) Subjects will be admitted in-house in the evening before the first study drug administration (Day 0) and will remain in-house for 24 and 36 hours after first (Day 1) and last (Day 10) doses, respectively; subjects will return for all other visits. PK blood samples will be drawn on Day 1 over 24 hours at designated time points as described below. Additionally, pre-dose (trough) samples will be drawn before dosing on Days 2, 3, 4, 5, 7, 8, and 9. On Day 10, blood samples will be collected over 36 hours at designated time points as described below and during additional visits at 48, 96, 120, 144, 168 and 192 hours post-dose. Subjects will be continuously monitored for safety. An End-of Study/Safety Follow-up visit will take place on the last PK sampling day, ie, 192 hours after the last dose administration.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male and female subjects, born in China, both parents of Chinese descent, aged at screening between 18-50 years old (inclusive), and having not lived outside of China for more than 10 years (in total, confirmed by verbal report).
2. BMI ≥ 18.0 and ≤ 30.0.
3. Subjects in general good health in the opinion of the investigator as determined by medical history, vital signs and physical examination.
4. No significant abnormalities in ECG (eg, prolonged QTcF, prolonged PR interval) done at screening and on Days (0) before dosing session.
5. No clinically significant abnormalities in hematology, blood chemistry, or urinalysis lab tests at screening.
6. No known history of alcohol or drug abuse. Subjects with negative urinary drugs of abuse (DOA) screen determined on Day (0) before dosing session(s).
7. Negative human immunodeficiency virus (HIV), hepatitis B, and hepatitis C serology tests as evaluated at screening.
8. Negative urine pregnancy tests at screening and at check-in (women of childbearing potential only).
9. . Subjects must be able to adhere to the visit schedule and protocol requirements and be available to complete the study.
10. All subjects must agree to use a highly effective method of birth control during the study and up to 15 days after the last study drug administration. A highly effective method of birth control is considered to be one of the following:

    * An oral or implanted hormonal method of contraception (if it had been used for ≥3 months prior to study drug administration) while also using a barrier method (ie, condom or diaphragm)
    * A hormone or copper intrauterine device if it had been in place for ≥3 months prior to study drug administration (subjects using nonhormonal or copper intrauterine devices were also required to use a barrier method of contraception)
    * A vasectomized partner
    * Total abstinence is acceptable; however, the subject is required to use a highly effective method of contraception if the subject decides subsequently not to abstain
    * Periodic abstinence around ovulation is not considered acceptable
    * Women who are either surgically sterilized or postmenopausal (last menstrual period at least 1 year prior to the screening visit) are exempt from this requirement. If medical records are not available to document sterility, urine pregnancy testing will be performed at screening and check-in.
11. Subjects must provide written informed consent to participate in the study.

Exclusion Criteria:

1. Documented history or on-going symptoms of any gastrointestinal disorder involving motility, gastric acid or gastric emptying or malabsorption, including but not limited to, peptic ulcer disease, gastroesophageal reflux, dyspepsia, gastroparesis, chronic diarrhea, chronic constipation, gall bladder disease, pancreatitis, lactose intolerance and celiac disease.
2. History of esophageal, gastric, biliary, or intestinal surgery (excluding herniotomy and appendectomy which are not related to gastrointestinal disorders).
3. Known history of significant medical disorder, which in the investigator's judgment contraindicates administration of the study medications.
4. Any clinically significant abnormality upon physical examination or in the clinical laboratory tests at screening visit.
5. Use of any prescription or over-the-counter (OTC) medications, vitamins and herbal or dietary supplements within 14 days prior to dosing. Paracetamol or ibuprofen for symptomatic relief of pain is allowed until 24 hours prior to the study drug administration.
6. Subjects who have taken anticholinergic or other drugs known to affect gastrointestinal motility within 7 days prior to the first dosing.
7. Treatment with any drugs with known hepatic enzyme-inducing or inhibiting agents (eg, barbiturates, phenothiazines, cimetidine, carbamazepine) within 30 days prior to dosing.
8. Known clinically significant hypersensitivity and/or allergy to any drugs.
9. Subjects with recent significant change in body weight (±10% within 3 months of screening).
10. Any acute illness (eg, acute infection) within 48 hours prior to the first study drug administration, which is considered of significance by the Principal Investigator.
11. Participation in another clinical trial with drugs, received within 3 months prior to dosing (calculated from the previous study's last dosing date).
12. Female subjects who are pregnant or breastfeeding.
13. Subjects who donated blood in the three months or received blood or plasma derivatives in the six months preceding study drug administration.
14. Inability to fast or consume the food provided in the study (including any clinically significant known food allergies or food restrictions).
15. Subjects who are non-cooperative, unwilling or unable to communicate with the investigators and site staff (ie, language problem, poor mental development or impaired cerebral function).

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2016-05; Primary Completion 2016-09 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose.Part C: Dosing days 1-10
Area under the plasma concentration time curve (AUC) | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose.Part C: Dosing days 1-10.
Maximum plasma concentration (Cmax) | Part B: Day 1 and day 10
Area under the plasma concentration time curve (AUC) | Part C: Day 1 and Day 10

SECONDARY OUTCOMES:
Adverse Event (AE) Profile | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose. Part B:Dosing days 1-10
  Adverse Events records in patients file
Adverse Event (AE) Profile | Part B: Dosing days 1 and 2: pre-dose (within 60 min before first dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18 and 24 (before second dosing) hours after drug administration+ day 3-10
  Adverse Events records in patients file
Clinical Laboratory Safety Tests | Part A:Pre-dose (within 60 min before dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18, 24, 30, 36, 48(±60 min), 72 (±60 min), 96 (±60 min), 144 (±60 min) hours post-dose. Part B:Dosing days 1-10
  Blood Tests
Clinical Laboratory Safety Tests | Part B:Dosing days 1 and 2: pre-dose (within 60 min before first dosing), 1, 2, 3, 4, 5, 6, 8, 10, 12, 14, 18 and 24 (before second dosing) hours after drug administration+ day 3-10
  Blood Tests

CONTACTS AND LOCATIONS:
Locations (1):
- WCCT Global, LLC., Cypress, California, United States